CLINICAL TRIAL: NCT02228369
Title: A Phase I, Open-label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumour Activity of AZD3759 or AZD9291 in Patients With EGFR Mutation Positive Advanced Stage Non Small Cell Lung Cancer (NSCLC)
Brief Title: Oral Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors, AZD3759 or AZD9291, in Patients Who Have Advanced Non-Small Cell Lung Cancer
Acronym: BLOOM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6030C00001
Record Dates: First submitted 2014-08-20; First posted 2014-08-29 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: EGFR Mutation Positive Advanced Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer, EGFR, Tyrosine kinase inhibitor,EGFR mutation positive, Brain Metastasis, Leptomeningeal Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Meningeal Carcinomatosis | interventions — AZD3759; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily dose of AZD3759 (Experimental): Daily oral dose of AZD3759
  Interventions: Drug: AZD3759
- Daily Dose of AZD9291 (Experimental): Daily oral dose of AZD9291
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD3759 — Starting dose 50 mg, administered twice daily. If tolerated subsequent cohorts will test increasing doses of AZD3759, until a maximum tolerated dose or an effective dose is defined
  Arms: Daily dose of AZD3759
Drug: AZD9291 — AZD9291 160mg once daily
  Arms: Daily Dose of AZD9291

SUMMARY:
This is the first time in patient study to assess the safety, tolerability and preliminary efficacy of AZD3759 in patients with advanced Non Small Cell Lung Cancer (NSCLC) In this study, patients with Leptomeningeal Metastasis and Brain Metastasis may also be enrolled to assess the anti-tumour efficacy, safety, pharmacokinetics and potential biological activity of AZD9291

DETAILED DESCRIPTION:
A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumour Activity of AZD3759 or AZD9291 in Patients with EGFR Mutation Positive Advanced Stage Non Small Cell Lung Cancer (NSCLC) who failed standard treatment and developed brain or leptomeningeal diseases

ELIGIBILITY:
Inclusion Criteria:

1. Obtained written informed consent
2. Male or female aged at least 18 years. Aged at least 20 if Japanese.
3. Histologically or cytologically confirmed diagnosis of NSCLC with single activating EGFR mutations (L858R or Exon19Del).
4. Eastern Cooperative Oncology Group performance status of 0 to1. For LM patients, 0 to 2 is acceptable.
5. In Part A, prior treatment with at least one line of a single agent EGFR TKI and at least 1 line of chemotherapy.
6. In Part B-BM expansion, patients must have not received any EGFR TKI and have asymptomatic brain metastasis, either found during screening process which does not require local treatment in the opinion of the investigator or local treatment has been given (surgery or radiation), patient must be stable without corticosteroid and/or anti-convulsants treatment for at least 2 weeks before study enrollment. For Part B-LM expansion, patients who received previous EGFR TKI treatment must have stable extracranial disease;EGFR TKI treatment naïve patients can also be enrolled into AZD9291 cohorts, or AZD3759 cohorts if efficacy signal seen in Part A and agreed by Safety Review Committee.
7. For patients with neither LM nor measurable BM: At least one measurable extracranial lesion. For patients with measurable BM but without LM: at least one measurable intracranial lesion
8. For patients with LM: Confirmed diagnosis of LM by positive CSF cytology.
9. Male patients should be willing to use barrier contraception, i.e., condoms, until 3 months after last study drug is taken.
10. Females should agree to use adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential
11. In Part B-AZD9291 LM expansion (sub-cohort of T790M+ LM patients), patients must have central confirmation of T790M+ mutation status from a sample taken after documented progression on the last treatment administered prior to enrolling in the study. Patients must have received prior therapy with an EGFR TKI and may also have received additional lines of treatment. Stable extracranial disease is not required.

Exclusion Criteria:

1. For patients with LM and/or BM, CNS complications that require urgent neurosurgical intervention
2. For patient with LM, inability to undergo collection of CSF
3. Treatment with an EGFR TKI (e.g., erlotinib or gefitinib) within 8 days or approximately 5 x half-life, whichever is the longer, of the first dose of study treatment.
4. Any cytotoxic chemotherapy,or other anticancer drugs for the treatment of advanced NSCLC from a previous treatment regimen within 14 days of the first dose of study treatment
5. Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment with the exception of patients receiving radiation to more than 30% of the bone marrow which must be completed within 4 weeks of the first dose of study treatment.
6. Patients currently receiving (or unable to stop use at least 1 week prior to receiving the first dose of AZD3759/AZD9291) medications or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 3A4/5 and potential inhibitors of cytochrome P450 2C8 (for patients to be enrolled into AZD9291 cohorts only).
7. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
8. Known intracranial haemorrhage which is unrelated to tumour
9. Refractory nausea and vomiting if not controlled by supportive therapy, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD3759/AZD9291
10. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses
11. Inadequate bone marrow reserve or organ function
12. Clinically significant ECG abnormalities or any factors that increase the risk of corrected QT interval prolongation or risk of arrhythmic events
13. Prior history of whole brain radiotherapy (only applicable for AZD3759 BM expansion)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2017-08-19 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability (The number of patients with each AE by system organ class, preferred term and CTCAE grade) | From Informed consent until the end of the follow-up period which is defined as 28 days (+7 days) after study treatment is discontinued.
  Adverse events will be collected from Informed consent until the end of the follow-up period which is defined as 28 days (+7 days) after study treatment is discontinued.Physical exam (screening, single dosing day, Day 1 of every 3-week cycle of multiple dosing and treatment discontinuation). ECG and vital signs (screening, Day 1 and 2 of Cycle 0 for AZD3759 cohorts, Day 8 of Cycle 1 for AZD3759 cohorts, Day 1 of every 3-week cycle, treatment discontinuation, and if occurrence of any cardiac adverse event). Lab variables (screening, first dosing day, Day 1, 8 and 15 of multiple dosing, Day 1 of every 3-week cycle and treatment discontinuation). Eye exam (at screening and study drug discontinuation and upon occurrence of any visual AE). Echocardiogram or multigated radionuclide angiography (at screening,whenever necessary as clinically indicated throughout the study for AZD3759 cohorts.

SECONDARY OUTCOMES:
Plasma concentration of AZD3759 and metabolite and pharmacokinetics parameters after single dose of AZD3759(Cmax, tmax, terminal rate constant, half life, AUC, clearance, volume of distribution, mean residence time) | Cycle 0 Day 1 to 3 in Part A patients.
  The parent drug and N-demethylated metabolite in plasma samples will be analyzed: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, hour in Day 1; 24hour in Day 2 and 48hour in Day 3.
  AUC: Area Under Curve
Plasma,urine,cerebrospinal fluid concentration of AZD3759 and metabolite and pharmacokinetics parameters after multiple dosing(Cmax,ss, tmax,ss, Cmin,ss, AUCss, CLss/F). | Blood samples: Cycle 1 Day 8 and Cycle 3 Day 1 in all patients. Urine samples: 0-12h at Cycle 1 Day 8 in Part A. CSF samples: pre-dose of Cycle 1 Day 8 in BM; Pre-dose of Cycle 1 Day 8 and Cycle 3 Day 1 in LM
  The parent drug and N-demethylated metabolite in plasma samples from all patients will be analyzed: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12hour on Cycle 1 Day 8 and Cycle 3 Day 1 . The parent drug and N-demethylated metabolite in urine samples from Part A patients will be analyzed: 0-12h at Cycle 1 Day 8. The parent drug and N-demethylated metabolite in cerebrospinal fluid samples will be analyzed: pre-dose of Cycle 1 Day 8 in brain metastasis patients; pre-dose of Cycle 1 Day 8 and Cycle 3 Day 1 in leptomeningeal metastasis patients. AUCss: Area Under Curve Steady State CLss: Clearance Steady State
Plasma,urine, cerebrospinal fluid concentration of AZD3759 and metabolite and pharmacokinetics parameters after multiple dosing (extent of accumulation, renal clearance, time dependency of pharmacokinetics and amount of drug excreted) | Blood samples: Cycle 1 Day 8 and Cycle 3 Day 1 in all patients. Urine samples: 0-12h at Cycle 1 Day 8 in Part A patients. CSF samples: pre-dose of Cycle 1 Day 8 and Cycle 3 Day 1 in Part B patients .
  The parent drug and N-demethylated metabolite in plasma samples from all patients will be analyzed: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12hour on Cycle 1 Day 8 and Cycle 3 Day 1. The parent drug and N-demethylated metabolite in urine samples from Part A patients will be analyzed: 0-12h at Cycle 1 Day 8. The parent drug and N-demethylated metabolite in cerebrospinal fluid samples will be analyzed: pre-dose of Cycle 1 Day 8 in brain metastasis patients; pre-dose of Cycle 1 Day 8 and Cycle 3 Day 1 in leptomeningeal metastasis patients.
Plasma, cerebrospinal fluid concentration of AZD9291 and metabolite and pharmacokinetics parameters after multiple dose of AZD9291(Cmax,ss, tmax,ss, Cmin,ss, AUCss, CLss/F). | Blood samples: Cycle 1 Day 1, 8, 15 and Cycle 2 Day 1. Cerebrospinal fluid samples: pre-dose of Cycle 2 Day 1 and pre-dose of Cycle 3 Day 1.
  The parent drug and metabolites in plasma samples from all patients treated with AZD9291 will be analyzed: pre-dose of Cycle 1 Day 1, 8, 15; pre-dose, 1, 1.5, 2, 4, 6, 8, 10, 12, 24hour on Cycle 2 Day 1. The parent drug and metabolites in cerebrospinal fluid samples will be analyzed: pre-dose of Cycle 2 Day 1 in brain metastasis patients; pre-dose of Cycle 2 Day 1 and Cycle 3 Day 1 in leptomeningeal metastasis patients . AUCss: Area Under Curve Steady State CLss: Clearance Steady State
Plasma, cerebrospinal fluid concentration of AZD9291 and metabolites and pharmacokinetics parameters after multiple dosing (extent of accumulation, renal clearance, time dependency of pharmacokinetics and amount of drug excreted) | Blood samples: Cycle 1 Day 1, 8, 15 and Cycle 2 Day 1. Cerebrospinal fluid samples: pre-dose of Cycle 2 Day 1 and pre-dose of Cycle 3 Day 1.
  The parent drug and metabolites in plasma samples from all patients treated with AZD9291 will be analyzed: pre-dose of Cycle 1 Day 1, 8, 15; pre-dose, 1, 1.5, 2, 4, 6, 8, 10, 12, 24hour on Cycle 2 Day 1. The parent drug and metabolites in cerebrospinal fluid samples will be analyzed: pre-dose of Cycle 2 Day 1 in brain metastasis patients; pre-dose of Cycle 2 Day 1 and Cycle 3 Day 1 in leptomeningeal metastasis patients . AUCss: Area Under Curve Steady State CLss: Clearance Steady State
Overall survival follow up for all expansion patients | Every 6 weeks after the 28- day safety follow-up visit
  After 28-day follow-up visit, patients will be followed for overall survival via telephone every 6 weeks until death, lost to follow-up or consent withdrawal
4b-hydroxy cholesterol in Part B patients with BM | pre-dose of Cycle 0 Day 1 and Cycle 1 Day 15
  Blood collection at pre-dose of Cycle 0 Day 1 and Cycle 1 Day 15 to evaluate if AZD3759 affects 4b-hydroxy cholesterol which is an endogenous marker of CYP enzyme induction
The effect of food on the pharmacokinetics of a single dose of AZD3759 in plasma | Cycle 0 Day 1 to Day 4 in Part B patients with BM
  Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hour of Cycle 0 Day 1and Day 4; 24 hour of Cycle 0 Day 2 and Day 4.A Mixed Effects model with treatment (fed/fasted) and period as fixed effects and patient as a random effect will be used to compare AUC/Cmax in the fed state with AUC/Cmax in the fasted state.
Cerebrospinal fluid response rate for patients with LM and/or BM | Screening and every 6 weeks (relative to first dose of multiple dosing) until progression, expected average 6 months
  Cerebrospinal fluid collection at screening and every 6 weeks until progression to evaluate the cerebrospinal fluid response rate which is defined as the percentage of leptomeningeal metastasis patients who have at least one cerebrospinal fluid response (100% clearance of tumour cells from cerebrospinal
Changes from baseline in central nervous system symptoms (analyzed from QLQ-BN20) in patients with LM treated with AZD3759 /AZD9291 | Screening, Day 1 of every 3-week cycle and treatment discontinuation, expected average 6 months.
  Quality of life questionnaire-Brain Cancer 20 questionnaire completed by patients at screening, Day 1 of every 3-week cycle and treatment discontinuation. Use relevant symptom questions to evaluate improvement of central nervous system symptoms.
Changes from baseline in neurological exam in patients with LM treated with AZD3759 /AZD9291 | Screening, Day 1 of every 3-week cycle and treatment discontinuation, expected average 6 months.
  Neurological exam will be performed: screening, single dosing day, Day 1 of every 3-week cycle of multiple dosing and treatment discontinuation
Measurement of Objective Response Rate (ORR) | Screening within 28days of treatments start and then every 6 weeks ± 1week(relative to first dose of multiple dosing) until objective disease progression or withdrawal from study,expected average 6 months.
  ORR assessed through the number of patients who achieve a disease response (i.e. complete response or partial response) assessed according to modified RECIST 1.1 criteria for central nervous system disease, extracranial disease and overall disease
Measurement of Disease Control Rate (DCR) | Screening within 28days of treatments start and then every 6 weeks ± 1week(relative to first dose of multiple dosing) until objective disease progression or withdrawal from study,expected average 6 months.
  DCR assessed through the number of patients who achieve a best response of confirmed CR, confirmed PR or responding, or stable disease according to modified RECIST 1.1 criteria for central nervous system disease, extracranial disease, leptomeningeal disease and overall disease
Measurement of Response Rate (RR) | Screening within 28days of treatments start and then every 6 weeks ± 1week(relative to first dose of multiple dosing) until objective disease progression or withdrawal from study,expected average 6 months.
  RR assessed through the number of patients who have at least one confirmed response of Complete Response or Responding prior to any evidence of progression according to modified RECIST 1.1 criteria for leptomeningeal disease
Measurement of Progression Free Survival (PFS) | Screening within 28days of treatments start and then every 6 weeks ± 1week(relative to first dose of multiple dosing) until objective disease progression or withdrawal from study,expected average 6 months.
  PFS assessed through change in tumour size (as well as assessment of non-target lesions and appearance of any new lesions) according to modified RECIST 1.1 criteria for Part B patients with brain metastasis and patients with leptomeningeal metastasis
Best Leptomeningeal Metastasis (LM) assessment for AZD9291 LM patients | Screening within 28days
  Best LM assessment via LANO criteria through the number of patients with LM present at baseline, without a requirement for confirmation. LANO assessments will be mapped to RECIST-like scores and performed via central imaging reading.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Yang, M.D. PhD, Study Director — Building 2, 199 Liangjing Road, Zhangjiang Hi-tech Park, Shanghai 201203, China
Locations (7):
- United States (2):
  - Research Site, Los Angeles, California
  - Research Site, Santa Monica, California
- Australia (2):
  - Research Site, Camperdown
  - Research Site, Heidelberg
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Research Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Yang JCH, Kim SW, Kim DW, Lee JS, Cho BC, Ahn JS, Lee DH, Kim TM, Goldman JW, Natale RB, Brown AP, Collins B, Chmielecki J, Vishwanathan K, Mendoza-Naranjo A, Ahn MJ. Osimertinib in Patients With Epidermal Growth Factor Receptor Mutation-Positive Non-Small-Cell Lung Cancer and Leptomeningeal Metastases: The BLOOM Study. J Clin Oncol. 2020 Feb 20;38(6):538-547. doi: 10.1200/JCO.19.00457. Epub 2019 Dec 6. PMID 31809241
- [Derived] Ahn MJ, Kim DW, Cho BC, Kim SW, Lee JS, Ahn JS, Kim TM, Lin CC, Kim HR, John T, Kao S, Goldman JW, Su WC, Natale R, Rabbie S, Harrop B, Overend P, Yang Z, Yang JC. Activity and safety of AZD3759 in EGFR-mutant non-small-cell lung cancer with CNS metastases (BLOOM): a phase 1, open-label, dose-escalation and dose-expansion study. Lancet Respir Med. 2017 Nov;5(11):891-902. doi: 10.1016/S2213-2600(17)30378-8. Epub 2017 Oct 19. PMID 29056570
- See also: BLOOM CSP_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2978&filename=BLOOM%20CSP_Redacted%20new.pdf
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search